CLINICAL TRIAL: NCT05682014
Title: The Effect of Web-Based Mindful Breastfeeding Program During Pregnancy on Postpartum Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Özge Şiir Dağlar, PhD student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IUC-OSDaglar-001
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Mindfulness; Breast Feeding; Psychological Well-Being
Keywords: Mindfulness; Breast Feeding; Psychological Well-Being
MeSH Terms: conditions — Breast Feeding; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Random sampling method will be used in the research. Randomization Pregnant women will be evaluated in terms of their eligibility for the study, a list of pregnant women included in the study will be created and divided into two groups. The assignment of pregnant women to the intervention and control groups in the study will be realized by assigning a number to each of the participants, forming a number group for the intervention group, and planning the numbers outside of this group as the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): A web-based "Mindful Breastfeeding Program", which is applied to pregnant women in groups of 5, consisting of 8 sessions, 2 sessions per week for 4 weeks.
  Mindful breastfeeding program will consist of breastfeeding education, introduction to the concept of mindfulness, mindful breastfeeding, practical suggestions to pregnant women by the researcher, providing a discussion environment for them to share their experiences, and homework on the content of the program.
  A web site with written material, video and audio recordings will be created and presented to the participants as a support element.
  In order for them to use mindfulness practices in their daily lives, motivational WhatsApp short messages will be sent by the researcher daily during the training, weekly during the post-training period, and daily in the postpartum period.
  Interventions: Behavioral: Mindful Breastfeeding Program
- Control Group (No Intervention): Only one session online breastfeeding training will be given and the training brochure for this training will be delivered to the participants via whatsapp.

INTERVENTIONS:
Behavioral: Mindful Breastfeeding Program — A web-based "Mindful Breastfeeding Program", which is applied to pregnant women in groups of 5, consisting of 8 sessions, 2 sessions per week for 4 weeks.
  Mindful breastfeeding program will consist of breastfeeding education, introduction to the concept of mindfulness, mindful breastfeeding, practical suggestions to pregnant women by the researcher, providing a discussion environment for them to share their experiences, and homework on the content of the program.
  A web site with written material, video and audio recordings will be created and presented to the participants as a support element.
  In order for them to use mindfulness practices in their daily lives, motivational WhatsApp short messages will be sent by the researcher daily during the training, weekly during the post-training period, and daily in the postpartum period.
  Arms: İntervention Group

SUMMARY:
The aim of this study is to evaluate the effectiveness of a web-based mindful breastfeeding program in pregnancy to increase awareness, breastfeeding adaptation and breastfeeding self-efficacy in postpartum breastfeeding. The Mindful breastfeeding program intervention will be compared to the group receiving basic breastfeeding education. The main hypothesis is that pregnant women included in the mindful breastfeeding program have higher postpartum breastfeeding awareness, breastfeeding adaptation and breastfeeding self-efficacy.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness of a web-based mindful breastfeeding program in pregnancy to increase awareness, breastfeeding adaptation and breastfeeding self-efficacy in postpartum breastfeeding.

There will be two groups in the study:

The web-based "Mindful Breastfeeding Program" (mindfulness-based breastfeeding program) consisting of 8 sessions in total, 2 sessions per week for 4 weeks, will be applied to the pregnant women who make up the intervention group. During the research, a QR code supported website will be established in order to support the awareness practices of the participants at home. While doing mindfulness practices at home, participants will be able to benefit from the short training videos on the website or the audio recordings prepared by the researcher with his own voice.

Only one session online breastfeeding training will be given to the control group and the training brochure for this training will be delivered to the participants via whatsapp.

A total of 40 pregnant women, 20 in the intervention group and 20 in the control group, will form the sample of the study. The main hypothesis is that the postpartum breastfeeding awareness, breastfeeding adaptation and breastfeeding self-efficacy of pregnant women included in the mindful breastfeeding program is higher than the pregnant women who participated in the single-session basic breastfeeding training.

Statistical analysis of the data obtained from the research will be made using SPSS (Statistical Packet for Social Science) for Windows 25.0 program.

ELIGIBILITY:
Inclusion Criteria for Research

* Able to communicate in Turkish,
* Being literate,
* Over 18 years old,
* Having primigravida,
* Conceiving naturally,
* Gestational week between 28-32 weeks,
* Having a single baby (no multiple pregnancy),
* Intention to breastfeed their baby after birth,
* The mother and her baby do not have any health problems,
* Having a smart phone and wireless internet,
* All pregnant women who score below 5 points in the depression sub-dimension, below 4 points in the anxiety sub-dimension, and below 8 points in the stress sub-dimension according to DASS-21 will be included in the sample.

Exclusion Criteria

* If the participant states that he/she wants to withdraw from the research,
* Not attending at least two training sessions,
* Premature birth (before 37 weeks of pregnancy),
* Not breastfeeding the baby after birth,
* Not participating in the post-test,
* Failure to complete the follow-up period for any reason.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Mindful Breastfeeding Scale | Mindful breastfeeding program at 1 month postpartum in intervention group and control group.
Breast Feeding Adaptation Scale | Mindful breastfeeding program at 1 month postpartum in intervention group and control group.
Postpartum Breastfeeding Self-Efficacy Scale | Mindful breastfeeding program at 1 month postpartum in intervention group and control group.

SECONDARY OUTCOMES:
Sociodemographic Information Form | Mindful breastfeeding program pre-intervention in intervention group and control group.
Antenatal Breastfeeding Self-Efficacy Scale | Mindful breastfeeding program pre-intervention in intervention group and control group.
Depression, Anxiety, Stress Scale | Mindful breastfeeding program pre-intervention in intervention group and control group.
Depression, Anxiety, Stress Scale | Mindful breastfeeding program at 1 month postpartum in intervention group and control group.
Mindfulness Scale | Mindful breastfeeding program pre-intervention in intervention group and control group.
Mindfulness Scale | Mindful breastfeeding program at 1 month postpartum in intervention group and control group.
Postpartum Breastfeeding Evaluation Form | Mindful breastfeeding program within the first 7 days postpartum in the intervention group and control group.
  A form developed by the researcher to evaluate the breastfeeding status of mothers in the first 7 days after birth (average between 3-5 days).
System Usability Scale | Immediately after intervention in the Mindful breastfeeding program intervention group.
  The usability of the website will be evaluated by the participants in the intervention group at the last session of the training program using the System Usability Scale (SUS).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No